CLINICAL TRIAL: NCT04924751
Title: National Taiwan University Hospital
Brief Title: Contrast-Enhanced Harmonic vs Conventional EUS-guided Fine Needle Biopsy for Solid Pancreatic Lesions: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201905065RIND
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Solid Lesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: At the time of the procedure, the endoscopy nurse opened an envelope containing computer-generated randomization assignments for the study patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEH-EUS-guided FNB group (Experimental): In CEH-EUS-guided FNB group, needle puncture directly to the enhancing area 15-20 times without passing to the non-enhancing area was performed. After each pass, the needle is removed and the stylet will be introduced into the needle to extrude any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). The total length of the MVC will be measured before placement into a formalin bottle. EUS-FNB is completed if the obtained MVC is longer than 4mm and deemed adequate by endoscopist. If the obtained MVC is < 4mm, the procedure is repeated until a MVC of ≥ 4mm is obtained and deemed adequate by endoscopist. A maximum of 7 passes is allowed.
  Interventions: Diagnostic Test: Endoscopic ultrasound-guided fine needle biopsy
- Conventional-EUS-guided FNB with fanning technique group (Active Comparator): In conventional-EUS-guided FNB with fanning technique group, the needle was positioned at four different areas within the mass and then moved back and forth four times in each area to procure tissue (4 × 4). After each pass, the needle is removed and the stylet will be introduced into the needle to extrude any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). The total length of the MVC will be measured before placement into a formalin bottle. EUS-FNB is completed if the obtained MVC is longer than 4mm and deemed adequate by endoscopist. If the obtained MVC is < 4mm, the procedure is repeated until a MVC of ≥ 4mm is obtained and deemed adequate by endoscopist. A maximum of 7 passes is allowed.
  Interventions: Diagnostic Test: Endoscopic ultrasound-guided fine needle biopsy

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound-guided fine needle biopsy — Under endoscopic ultrasound guidance, fine-needle biopsy is used to collect biopsy samples from solid pancreatic lesions throughout the digestive tract and is useful in diagnosing solid pancreatic lesions.

SUMMARY:
In the previous studies, EUS-guided fine needle aspiration (FNA) with fanning technique in solid pancreatic lesions (SPLs) with avascular areas had a negative impact on diagnostic accuracy of FNA. Because of the retrospective basis of previous studies, a prospective study is warranted to answer whether contrast-enhanced harmonic(CEH) EUS-guided FNA/B is superior to conventional EUS-guided FNA/B with fanning technique in SPLs. The main objective of this randomized trial therefore was to determine whether CEH-EUS-guided sampling to avoid non-enhanced areas within a mass lesion result in more rapid diagnosis requiring fewer FNB passes than the conventional EUS-guided FNB with fanning needle throughout the mass is targeted.

DETAILED DESCRIPTION:
A prospective randomized controlled study was undertaken of patients with solid pancreatic mass lesions who were referred for EUS. Total 120 patients were randomized with 1:1 ratio into undergo CEH-EUS-guided FNB or conventional EUS-guided FNB with fanning technique. At the time of the procedure, the endoscopy nurse opened an envelope containing computer-generated randomization assignments for the study patients. All procedures were performed by a linear array echoendoscope (Olympus UCT260; Olympus, Tokyo, Japan). Procedures were performed under conscious sedation with patients in the left lateral decubitus position.

In CEH-EUS-guided FNB group, needle puncture directly to the enhancing area 15-20 times without passing to the non-enhancing area was performed. In conventional-EUS-guided FNB with fanning technique group, the needle was positioned at four different areas within the mass and then moved back and forth four times in each area to procure tissue (4 × 4). After each pass, the needle is removed and the stylet will be introduced into the needle to extrude any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). The total length of the MVC will be measured before placement into a formalin bottle. EUS-FNB is completed if the obtained MVC is longer than 4mm and deemed adequate by endoscopist. If the obtained MVC is < 4mm, the procedure is repeated until a MVC of ≥ 4mm is obtained and deemed adequate by endoscopist. A maximum of 7 passes is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 20years, referred for EUS-guided tissue acquisition for solid pancreatic lesions greater than 1cm in the largest diameter will be recruited.

Exclusion Criteria:

* Patients with coagulopathy, altered anatomy, contraindications for conscious sedation, pregnancy and those who cannot provide informed consent would be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-03-17 (Estimated)

PRIMARY OUTCOMES:
the median number of passes required to establish a diagnosis | 1 day
  EUS-FNB is completed if the obtained macroscopic visible core (MVC) is longer than 4mm and deemed adequate by endoscopist

SECONDARY OUTCOMES:
diagnostic accuracy rate | 3 months
  Diagnostic accuracy was defined as the proportion of patients in whom successful diagnosis was reached within the procedure
overall complication rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided